CLINICAL TRIAL: NCT07149324
Title: Can a Single Session Intervention Decrease Eating Disorder Symptoms in At-risk University Students? A Pilot Study.
Brief Title: Can a Single-session Intervention Decrease Risk for Mental Health Symptoms in Young Adults? A Preliminary Investigation of Feasibility and Acceptability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chloe White (Other)
Responsible Party: Sponsor-Investigator, Chloe White, Project Director, Simon Fraser University
Organization: Simon Fraser University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 518585
Record Dates: First submitted 2025-07-23; First posted 2025-09-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Disordered Eating Behaviors; Disordered Eating
Keywords: Eating disorders; Depression; Self-esteem
MeSH Terms: conditions — Disordered Eating Behavior; Feeding and Eating Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This will be a case series study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Other)
  Interventions: Behavioral: Single Session for Overevaluation

INTERVENTIONS:
Behavioral: Single Session for Overevaluation — A single session informed by the principles of Cognitive Behavioural Therapy-Enhanced and motivational intervening.

SUMMARY:
This project has two primary aims: 1) to develop a single session intervention to understand different forms of self-evaluation with input from young adults, and 2) to examine whether a single session can improve the ways in which young adults measure their self-importance with a session led by a trained masters-level therapist. Eligible participants will complete a baseline questionnaire, a therapeutic session online, and follow-up questionnaires.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of the present study is to 1) seek input from young adults regarding the utility, content and structure of a single session intervention, and 2) to examine whether a single session can alter mental health symptoms in young adults. Specifically, the study will seek to examine how intervening with a core risk factor of disordered eating and low mood, self-evaluation based in appearance, may influence mental health symptoms, including self-esteem, low mood, disordered eating, and body satisfaction.

JUSTIFICATION:

This study is important for various reasons. Basing one's self-esteem nearly exclusively on appearance-related variables (e.g., shape, weight) is a risk factor for negative mental health symptoms, such as disordered eating, low mood, and diminished self-esteem. Thus, self-esteem based on appearance may be an important place to intervene to decrease potential negative mental health outcomes and increase resiliency. However, interventions which are designed to treat over reliance on appearance in evaluating one's self-esteem range between 16-20 sessions in duration and are often time and cost inefficient to provide to all individuals who evaluate themselves based on their appearance; and importantly, single session interventions have been shown to increase mood, healthy eating behaviours, and body satisfaction in young adults and adolescents. Thus, there exists a need for highly specific and specialized interventions which are informed by known past risk factors, such as overevaluation of appearance. Thus, development and testing of a single session intervention developed through consideration of research on interventions for disordered eating, low mood, and diminished self-esteem to date, and through consult with overevaluation of appearance, is a critical development to diminish the overall negative health consequences of a dysfunctional system of self-evaluation.

Given the paucity of research conducted on this specific topic to date, the present study will conduct two phases of the same study to examine a novel single session intervention to change how participants measure their self-importance. A checklist outlining the various components of the intervention session is in the Support Documents section. In brief, the intervention session will begin with individuals completing a modified version of the Shape and Weight-Based Self-Esteem Inventory (SAWBS) to assess their self-reliance on (overevaluation of) appearance. After completing this measure, participants and the clinician will discuss the participants overevaluation in reference to the average levels of overevaluation of other individuals their age. Additionally, the clinician will provide psychoeducation about their overevaluation in reference to the individual's risk for negative mental health outcomes (e.g., low mood, disordered eating, anxiety). Importantly, discussions and psychoeducation will be tailored by the therapist to intervene specifically with symptoms that are identified as the most concerning by the participant. Following this discussion, participants will complete a reflective writing exercise, complete the SAWBS again indicating which areas bring them pleasure that they would like to increase, and come up with a plan of action to enhance reliance on other areas that are important to them.

Recruitment will occur in two phases. Phase I will be focused on intervention development. In Phase I, five eligible participants will receive the intervention session, followed by two brief interviews designed to gather feedback about the intervention session. Importantly, these interviews will be led by trained research assistants who have completed masters in Clinical Psychology rather than the lead therapist. In these interviews, participants will be asked about their experience of the session, whether they would change anything about the session, their preference for duration or structure of the session, and will be provided with open-ended opportunities to discuss anything else relevant to their experience in the study. They will also complete a secondary interview one week following the intervention, which will include open-ended questions about the efficacy of the session over the past week and provide them with a second opportunity to provide feedback about the session content. This phase will also include a series of measures completed at pre-intervention, including demographic questions. Additionally, some measures will be completed at post-intervention (measures in Supported Documents). The measures completed will be a well-validated measure of disordered eating symptoms (the Eating Disorder-15), select questions from the Eating Disorder Examination-Questionnaire (EDE-Q), a measure of overevaluation of appearance (Shape and Weight Based Self-Esteem Inventory), a quantitative measure of session acceptability (Program Feedback Scale), a measure of body satisfaction (BSS; ), and a measure of mood (BHS-4). Importantly, adequate acceptability of the intervention, demonstrated via responses on the Program Feedback Scale of equal to or >3.5/5, and qualitative interviews (interview questions provided in Supported Documents) will need to be demonstrated across participants to proceed with Phase II.

Phase II will be a case series study, with the goal of examining the utility of the single session intervention at modifying how participants measure their self-importance over a four-week period. A case series will be used to capitalize on the relatively rare population of individuals with demonstrated heightened overvaluation of appearance. Additionally, a case series study will allow researchers to develop increasingly fine-grained hypotheses about the feasibility of a single session intervention for intervening with over reliance on appearance in self-evaluation, a presently unknown possibility. In Phase II, ten eligible participants will receive the intervention session, followed by two brief follow-up questionnaires. These participants will complete a pre-intervention questionnaire, a post-intervention questionnaire, a one-week follow-up questionnaire, and a four-week follow-up questionnaire. In the pre-intervention questionnaire, participants will provide demographic information and will complete a well-validated measure of disordered eating (the Eating Disorder-15), select questions from the Eating Disorder Examination-Questionnaire (EDE-Q), as well as measures of overevaluation of appearance (Shape and Weight Based Self-Esteem Inventory), body shape satisfaction, and low mood. In the post-intervention questionnaire, they will complete the body shape satisfaction scale, select questions from the Eating Disorder Examination-Questionnaire (EDE-Q), the measure of mood (BHS-4), and a measure of session acceptability (Program Feedback Scale, PFS). The one-week follow-up will include the measure of disordered eating symptoms (ED-15 & EDE-Q), body shape satisfaction, and the measure of mood. The four-week follow-up will include the measure of disordered eating, body shape satisfaction, mood, and overevaluation of appearance. Each participant will be prompted to respond to 1- and 4-week follow-up questionnaires via their preferred method of contact (email or text message).

STATISTICAL ANALYSES:

Statistical analyses will be descriptive in nature given the treatment development and case series design. These designs do not require large sample sizes and increase focus on patterns within participants, rather than between. Thus, inferential statistics are not used and no apriori power analyses were conducted. Alternatively, to determine sample size, a careful surveillance of literature on case series studies and treatment development was undertaken. Analyses for Phase I will include examining the qualitative feedback given by the five participants regarding the session content for themes and examination of the Program Feedback Scale item-level responses across participants through measures of central tendency (e.g., mean). Analyses for Phase II will examine trends of the ten participant scores across measures using measures of central tendency and plotting various data points on graphs. All measures, including mood, disordered eating, overevaluation, body shape satisfaction, and the program feedback scale will be examined using these techniques for all participants.

ELIGIBILITY:
Inclusion Criteria:

* between 18-25 years of age
* English speaking
* Demonstrate elevated overevaluation of weight, shape or muscularity

Exclusion Criteria:

* Have or have had in the past an eating disorder
* Is receiving treatment for an eating disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Shape and Weight Based Self-Esteem Inventory (SAWBS) | From enrollment to the end of follow-up at 4-weeks
  Pie graph between 0-100. Higher scores indicate greater overevaluation of shape, weight or muscularity.
Eating Disorder-15 (ED-15) | From enrollment to the end of follow-up at 4-weeks
  The ED-15 is comprised of 15 questions and uses a 7-point rating scale (0 - 6) for each item, with higher scores suggesting a greater likelihood or presence of eating disorder symptoms.
Eating Disorder Examination - Questionnaire (EDE-Q) | From enrollment to the end of follow-up at 4-weeks
  The EDE-Q is comprised of 28 questions and uses a 7-point rating scale (0-6) for each item, with higher scores reflecting greater ED symptoms.
Program Feedback Scale (PFS) | Immediately after the intervention
  The PFS is a 9-item questionnaire which was developed to examine acceptability of SSI's. Items one through seven are rated on a 5-point Likert-type scales ranging from 0 (really disagree) to 4 (really agree). Higher scores indicate greater acceptability of the single session. The remaining two items are open-ended questions (e.g., "What did you like about the program?") which allow for participants to provide detailed feedback.

SECONDARY OUTCOMES:
Beck Hopelessness Scale-4 (BHS-4) | From enrollment to the end of follow-up at 4-weeks
  The BHS-4 is a 4-item measure asking participants to rate their sense of hopelessness using a 4-item Likert-type scale. A total score is formed from summing across all 4-items to form an overall total score which signifies the extent to which the individual is experiencing hopelessness; thus, a higher score indicates greater depressive symptoms.
Body Shape Satisfaction Scale - 10 (BSS-10) | From enrollment to the end of treatment at 4-weeks
  The Body Shape Satisfaction Scale - 10 is an abbreviated version of the Body Shape Satisfaction Scale. The 10-item questionnaire uses a 5-point Likert type scale, ranging from 1 (very dissatisfied) to 5 (very satisfied), to indicate the extent to which participants are satisfied with different parts of their bodies. Higher scores indicate greater satisfaction with different body parts.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Zaitsoff, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data of measures used in the study will be shared.
Supporting Information: SAP, Analytic Code
Time Frame: The IPD will be available only after data analyses have concluded. Thus, an approximate date is in 2028

REFERENCES:
- [Background] White C, Maraun M, Zaitsoff S. How do I evaluate myself? The importance of examining overevaluation of muscularity in risk for eating disorder symptoms. J Eat Disord. 2025 Oct 23;13(1):233. doi: 10.1186/s40337-025-01419-3. PMID 41131650
- See also: Online SAWBS — https://gleaming-brioche-43ce26.netlify.app